CLINICAL TRIAL: NCT06517901
Title: MRI-targeted Fusion or Cognitive Ultrasound-guided Biopsy to Detect Prostate Cancer
Brief Title: Fusion or Cognitive Ultrasound-guided Biopsy to Detect Prostate Cancer
Acronym: FOCUS-PC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 7028
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer; Diagnosis
Keywords: Prostate; Cancer; Biopsy; Diagnosis; MRI
MeSH Terms: conditions — Prostatic Neoplasms; Disease; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Software fusion biopsy (Active Comparator): Software fusion biopsy: Biopsy of the MRI-detected lesion using an image fusion platform such as UroNav or similar.
  Interventions: Procedure: Software fusion prostate biopsy
- Cognitive fusion biopy (Experimental): Cognitive fusion biopsy: Biopsy of the MRI-detected lesion using visual estimation and/or measurements to identify landmarks and lesions.
  Interventions: Procedure: Cognitive fusion prostate biopsy

INTERVENTIONS:
Procedure: Software fusion prostate biopsy — Software fusion biopsy: Each participant in this study arm will first undergo biopsy of the MRI-detected lesion using an image fusion platform such as UroNav or similar. Three biopsy cores will be taken per lesion, with a maximum of three lesions being sampled per participant. Then systematic samples will be taken from the remainder of the prostate as per standard protocol (10-12 cores).
  Arms: Software fusion biopsy
Procedure: Cognitive fusion prostate biopsy — Cognitive fusion biopsy: Each participant in this study arm will first undergo biopsy of the MRI-detected lesion using visual estimation and/or measurements of lesion. Three biopsy cores will be taken per lesion, with a maximum of three lesions being sampled per participant. Then systematic samples will be taken from the remainder of the prostate as per standard protocol (10-12 cores).
  Other Names: Visual estimation fusion prostate biopsy
  Arms: Cognitive fusion biopy

SUMMARY:
The MRI-targeted biopsy for prostate cancer detection can be performed using one of two techniques:

1. Software-based fusion of MRI and ultrasound images (software fusion) or
2. Visually estimated MRI-informed (cognitive fusion) technique

To date, there is a lack of adequately powered RCTs directly comparing the cognitive vs fusion targeted biopsy. This randomized study will directly compare the detection rates of clinically significant prostate cancer following either the cognitive or the fusion targeted prostate biopsy in men with suspicious lesions noted on multi-parametric MRI (mp-MRI) of prostate.

DETAILED DESCRIPTION:
For prostate cancer detection, pre-biopsy multi-parametric magnetic resonance imaging (mp-MRI) followed by MRI-targeted prostate biopsy is standard of care which is supported by the guidelines from the American Urological Association and the European Association of Urology. The MRI-targeted prostate biopsy is associated with a significant increase in the detection of clinically significant prostate cancer (csPCa) compared to the ultrasound guided biopsy. The MRI-targeted biopsy can be performed using one of two techniques including software-based fusion of MRI and ultrasound images (software fusion) or visually guided MRI-informed (cognitive fusion) technique.

With regards to the diagnostic performance in detecting csPCa, current literature does not demonstrate a clear advantage to one targeting technique over the other. A systematic review and meta-analysis (published in early 2024) by Falagario et al evaluated all of the comparative studies of the above-mentioned MRI-targeting techniques. Of the 20 studies included, six reported improved detection of csPCa with fusion technique, one reported an advantage to the cognitive technique, while thirteen reported no significant difference. Of note, the majority of the studies were retrospective, with high risk of bias, that lacked uniform definition of csPCa, and employed variable mp-MRI technique (1.5T vs 3T) and scoring system (Likert vs PIRADS). There were only three small, prospective, randomized studies (RCT) available in the systematic review of literature. One RCT reported the fusion technique to be superior while two demonstrated no difference in csPCa detection rates. There was no significant difference in the detection of csPCa between the targeting techniques, however, low quality of evidence and heterogeneity warranted well-designed prospective studies.

Other studies, as well as personal experience, point to somewhat improved cancer detection the cognitive MRI-targeting approach, although the rates may be affected by patient selection related to lesion size and location.

Thus, the investigators are conducting an RCT to direct compare the csPCa detection rates following either the cognitive or the fusion targeted prostate biopsy in men with suspicious lesions noted on mp-MRI of prostate. The investigators hypothesize that the diagnostic accuracy MRI-targeted prostate biopsy using cognitive fusion technique is either similar to or not significantly inferior to the software fusion technique.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing prostate biopsy (either transrectal or transperineal) for suspected prostate cancer as part of their regular medical care
* Must be eligible to undergo both prostate biopsy procedure (cognitive or fusion)
* Men undergoing their first prostate biopsy procedure or with no previous prostate biopsy within 3 years
* Pre-biopsy mp-MRI of prostate with one or more lesions classified as PIRADS 3-5
* Largest dimension of any lesion on mp-MRI to be ≤ 2 cm
* Prostate-specific antigen level ≤ 20 ng/mL and/or abnormal digital rectal examination

Exclusion Criteria:

* mp-MRI detected lesions that are > 2 cm
* History of prostate biopsy within 3 years
* Previous diagnosis of prostate cancer
* Contraindications to prostate biopsy (eg, fever, evidence of genito-urinary infection, excessive co-morbidities as per treating physician)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1306 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Detection of clinically significant prostate cancer | 1 year
  Compare the overall detection of clinically significant prostate cancer following fusion vs cognitive MRI-targeted biopsy

SECONDARY OUTCOMES:
Detection of clinically significant prostate cancer in the targeted cores, systematic biopsy cores, and combined | 1 year
  Compare the detection of prostate cancer following fusion vs cognitive MRI-targeted biopsy
Detection of clinically significant prostate cancer based on lesion size (< 0.5 cm; 0.5 cm to 1 cm; > 1.1 cm etc) | 1 year
  Compare the detection of prostate cancer following fusion vs cognitive MRI-targeted biopsy
Detection of clinically significant prostate cancer at various lesion location (anterior, posterior, apex, base) | 1 year
  Compare the detection of prostate cancer following fusion vs cognitive MRI-targeted biopsy
Detection rate of overall prostate cancer of any grade | 1 year
  Compare the detection of prostate cancer following fusion vs cognitive MRI-targeted biopsy
Detection rate of clinically insignificant (low grade) prostate cancer | 1 year
  Compare the detection of prostate cancer following fusion vs cognitive MRI-targeted biopsy
Detection rate of clinically significant prostate cancer based on PSA density (PSA level / prostate volume) | 1 year
  Compare the detection of prostate cancer following fusion vs cognitive MRI-targeted biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Badar M Mian, MD, Study Chair — Albany Medical College
Locations (4):
- United States (3):
  - Lahey Clinic, Inc, Burlington, Massachusetts
  - Albany Medical Center, Albany, New York
  - Pennsylvania State University, Hershey, Pennsylvania
- Manitoba Prostate Centre, CancerCare Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Siddiqui MM, Rais-Bahrami S, Turkbey B, George AK, Rothwax J, Shakir N, Okoro C, Raskolnikov D, Parnes HL, Linehan WM, Merino MJ, Simon RM, Choyke PL, Wood BJ, Pinto PA. Comparison of MR/ultrasound fusion-guided biopsy with ultrasound-guided biopsy for the diagnosis of prostate cancer. JAMA. 2015 Jan 27;313(4):390-7. doi: 10.1001/jama.2014.17942. PMID 25626035
- [Background] Falagario UG, Pellegrino F, Fanelli A, Guzzi F, Bartoletti R, Cash H, Pavlovich C, Emberton M, Carrieri G, Giannarini G. Prostate cancer detection and complications of MRI-targeted prostate biopsy using cognitive registration, software-assisted image fusion or in-bore guidance: a systematic review and meta-analysis of comparative studies. Prostate Cancer Prostatic Dis. 2025 Jun;28(2):270-279. doi: 10.1038/s41391-024-00827-x. Epub 2024 Apr 5. PMID 38580833
- [Background] Izadpanahi MH, Elahian A, Gholipour F, Khorrami MH, Zargham M, Mohammadi Sichani M, Alizadeh F, Khorrami F. Diagnostic yield of fusion magnetic resonance-guided prostate biopsy versus cognitive-guided biopsy in biopsy-naive patients: a head-to-head randomized controlled trial. Prostate Cancer Prostatic Dis. 2021 Dec;24(4):1103-1109. doi: 10.1038/s41391-021-00366-9. Epub 2021 Apr 27. PMID 33907293
- [Background] Arsov C, Rabenalt R, Blondin D, Quentin M, Hiester A, Godehardt E, Gabbert HE, Becker N, Antoch G, Albers P, Schimmoller L. Prospective randomized trial comparing magnetic resonance imaging (MRI)-guided in-bore biopsy to MRI-ultrasound fusion and transrectal ultrasound-guided prostate biopsy in patients with prior negative biopsies. Eur Urol. 2015 Oct;68(4):713-20. doi: 10.1016/j.eururo.2015.06.008. Epub 2015 Jun 23. PMID 26116294
- [Background] Wegelin O, Exterkate L, van der Leest M, Kummer JA, Vreuls W, de Bruin PC, Bosch JLHR, Barentsz JO, Somford DM, van Melick HHE. The FUTURE Trial: A Multicenter Randomised Controlled Trial on Target Biopsy Techniques Based on Magnetic Resonance Imaging in the Diagnosis of Prostate Cancer in Patients with Prior Negative Biopsies. Eur Urol. 2019 Apr;75(4):582-590. doi: 10.1016/j.eururo.2018.11.040. Epub 2018 Dec 3. PMID 30522912
- [Background] Mian BM, Feustel PJ, Aziz A, Kaufman RP Jr, Bernstein A, Fisher HAG. Clinically Significant Prostate Cancer Detection Following Transrectal and Transperineal Biopsy: Results of the Prostate Biopsy Efficacy and Complications Randomized Clinical Trial. J Urol. 2024 Jul;212(1):21-31. doi: 10.1097/JU.0000000000003979. Epub 2024 May 3. PMID 38700844
- [Background] Hu JC, Assel M, Allaf ME, Ehdaie B, Vickers AJ, Cohen AJ, Ristau BT, Green DA, Han M, Rezaee ME, Pavlovich CP, Montgomery JS, Kowalczyk KJ, Ross AE, Kundu SD, Patel HD, Wang GJ, Graham JN, Shoag JE, Ghazi A, Singla N, Gorin MA, Schaeffer AJ, Schaeffer EM. Transperineal Versus Transrectal Magnetic Resonance Imaging-targeted and Systematic Prostate Biopsy to Prevent Infectious Complications: The PREVENT Randomized Trial. Eur Urol. 2024 Jul;86(1):61-68. doi: 10.1016/j.eururo.2023.12.015. Epub 2024 Jan 11. PMID 38212178
- [Background] Ploussard G, Barret E, Fiard G, Lenfant L, Malavaud B, Giannarini G, Almeras C, Aziza R, Renard-Penna R, Descotes JL, Rozet F, Beauval JB, Salin A, Roupret M. Transperineal Versus Transrectal Magnetic Resonance Imaging-targeted Biopsies for Prostate Cancer Diagnosis: Final Results of the Randomized PERFECT trial (CCAFU-PR1). Eur Urol Oncol. 2024 Oct;7(5):1080-1087. doi: 10.1016/j.euo.2024.01.019. Epub 2024 Feb 24. PMID 38403523
- [Background] Ortner G, Mavridis C, Fritz V, Schachtner J, Mamoulakis C, Nagele U, Tokas T. The Added Value of MRI-Based Targeted Biopsy in Biopsy-Naive Patients: A Propensity-Score Matched Comparison. J Clin Med. 2024 Feb 27;13(5):1355. doi: 10.3390/jcm13051355. PMID 38592166
- See also: American Urological Association guidelines — https://www.auanet.org/guidelines-and-quality/guidelines/early-detection-of-prostate-cancer-guidelines
- See also: European Association for Urology guidelines — https://uroweb.org/guidelines/prostate-cancer/chapter/diagnostic-evaluation